CLINICAL TRIAL: NCT04238611
Title: Minimally-Invasive Realtime Assessment of Continuous Lactate in Exercise
Acronym: MIRACLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 19HH5646
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Exercise; Lactate
Keywords: Minimally-invasive; Microneedle
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lactate microneedle (Experimental): Measurement of lactate through microneedle
  Interventions: Device: Microneedle; Diagnostic Test: Blood lactate measurement; Other: Exercise regimen

INTERVENTIONS:
Device: Microneedle — Lactate microneedle applied on the skin of participant
Diagnostic Test: Blood lactate measurement — Serum lactate testing through conventional laboratory methods
Other: Exercise regimen — Standardised aerobic exercise regimen

SUMMARY:
Lactate is a compound produced as a by-product of glycolysis. The increase in lactate concentration can result from a variety of causes, such as during anaerobic metabolism in exercise or haemodynamic shock in conditions such as sepsis.

The study will aim to validate a novel microneedle-based minimally invasive device for the continuous measurement of lactate during exercise.

DETAILED DESCRIPTION:
Lactate is a compound produced as a by-product of glycolysis. The increase in lactate concentration can result from a variety of causes, such as during anaerobic metabolism in exercise. The measurement of blood lactate during exercise has been routinely used to determine individual anaerobic thresholds, and optimise training in athletes.

The measurement of the lactate trend requires multiple blood tests, and this can be uncomfortable. The need for repeated procedures may therefore restrict the full utility of the biomarker. Although point-of-care lactate measurements are possible, the barriers to initiating testing may also limit its role in clinical decision-making.

The aim of the study is the validation of the microneedle-based lactate biosensor for real-time continuous lactate measurement in healthy volunteers during exercise as proof-of-concept.

ELIGIBILITY:
Inclusion Criteria:

1. Consenting adults ≥ 18 years old
2. Healthy with no other previous medical history
3. Able to perform moderately intensive exercise without difficulty for at least 30 minutes continuously, and engages in regular aerobic exercise at least twice a week

Exclusion Criteria:

1. Active inflammatory skin condition such as eczema or dermatitis
2. Active soft tissue infection or infection at any site
3. Known hypersensitivity to any microneedle component or dressings
4. Presence of any implantable electronic devices such as a pacemaker or stimulators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Performance of microneedle | 30 minutes
  Precision and accuracy of the lactate microneedle with reference to venous lactate as a gold standard. Current output from microneedle will be analysed against venous lactate and microdialysis lactate concentrations taken from participants every 5 minutes and concordance assessed through Bland-Altman analyses.

SECONDARY OUTCOMES:
Acceptability | 2 hours
  Participant acceptability of the biosensor through an end-of-study questionnaire in terms of pain, comfort, physical restriction and skin sensation using a visual analogue scale between 0 to 10 cm, where increased discomfort is represented by a higher score.

CONTACTS AND LOCATIONS:
Overall Officials: Alison H Holmes, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ming DK, Jangam S, Gowers SA, Wilson R, Freeman DM, Boutelle MG, Cass AE, O'Hare D, Holmes AH. Real-time continuous measurement of lactate through a minimally invasive microneedle patch: a phase I clinical study. BMJ Innov. 2022 Apr;8(2):87-94. doi: 10.1136/bmjinnov-2021-000864. Epub 2022 Feb 28. PMID 40979517